CLINICAL TRIAL: NCT07193706
Title: A Volume-Matched Quasi-Experimental Trial Comparing Micro-Dosed and Traditional Plyometric Training on Speed and Explosive Abilities in Elite Under-19 Soccer Players During the Pre-Season
Brief Title: Micro-Dosed vs. Traditional Plyometric Training in Elite Youth Soccer
Acronym: TRMD-PLYO_U19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matej Bel University (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Marián Škorik, PhD Candidate, Faculty of Sports Science and Health, Matej Bel University, Matej Bel University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 409/2024
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Plyometric Exercises; Soccer Performance; Speed; Explosive Strength; Microdosing
Keywords: Micro-dosed plyometric training; Youth soccer players; Explosive strength; Sprint performance; reactive strength

STUDY DESIGN:
Intervention Model Description: This is a parallel-group, quasi-experimental design. Players were allocated into two groups (micro-dosed vs. traditional plyometric training) using performance-based ranking (countermovement jump and drop jump tests) to achieve balanced groups. Both groups completed the similiar total weekly training volume during the 8-week pre-season period.
Masking Description: Masking was not feasible due to the visible differences in training frequency and scheduling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Plyometric Training Group (Active Comparator): Participants in this group completed a traditional plyometric training program during the 8-week pre-season period. The program consisted of 2 sessions per week, each lasting about 40 minutes. Exercises included countermovement jumps, drop jumps, broad jumps, and other standard plyometric drills. The total weekly training volume was matched to the micro-dosed group.
  Interventions: Behavioral: Traditional group training program
- Micro-dosed Plyometric Training Group (Experimental): Participants in this group completed a micro-dosed plyometric training program during the 8-week pre-season period. The program consisted of 3 to 4 shorter sessions per week, each lasting about 20 minutes. The same types of plyometric exercises were used as in the traditional group (e.g., countermovement jumps, drop jumps, broad jumps). The total weekly training volume was matched to the traditional group.
  Interventions: Behavioral: Micro-dosed group training program

INTERVENTIONS:
Behavioral: Traditional group training program — This intervention consists of two supervised plyometric training sessions per week, each lasting about 40 minutes. It represents the traditional approach with fewer but longer sessions. The total weekly training volume is equivalent to the micro-dosed group but distributed differently.
  Other Names: Traditional Group; TRG
  Arms: Traditional Plyometric Training Group
Behavioral: Micro-dosed group training program — This intervention consists of three to four shorter supervised plyometric sessions per week, each lasting about 20 minutes. It represents a micro-dosed approach, with higher frequency but shorter duration per session. The total weekly training volume is equivalent to the traditional group but distributed across more frequent sessions.
  Other Names: Micro-dose group; MDG
  Arms: Micro-dosed Plyometric Training Group

SUMMARY:
The goal of this clinical trial is to learn if a micro-dosed plyometric training program works as well as a traditional plyometric program for improving speed and explosive abilities in elite under-19 soccer players during the pre-season.

The main questions are:

1. Does micro-dosed training improve explosive and speed abilites, such as jumping and sprinting, as much as traditional training?
2. Does it improve reactivity and change-of-direction ability ?

Researchers will compare two groups:

* Traditional Training Group: 2 sessions per week, about 40 minutes each.
* Micro-dosed Group: 3-4 shorter sessions per week, about 20 minutes each. Both groups will complete the same total weekly training volume.

Participants will:

* Take part in an 8-week plyometric training program during pre-season.
* Complete performance tests (CM jump tests, a 30-meter sprint, and a 15-0-5 change-of-direction test, broad jump test, drop jump test) before and after 8-week plyometric intervention, .

This study will help coaches and players understand if shorter, more frequent plyometric training sessions can be a good alternative to traditional longer sessions when weekly training load is matched.

ELIGIBILITY:
Inclusion Criteria:

* Active membership in a U19 elite soccer club during the intervention.
* Medical fitness to participate in plyometric training and testing.
* Attendance at ≥75% of training sessions.
* Completion of all mandatory pre- and post-tests.
* Previous experience with plyometric training and testing procedures.

Exclusion Criteria:

* Medical limitations preventing safe participation in training or testing.
* Attendance lower than 75% of scheduled intervention sessions.
* Failure to complete mandatory baseline or follow-up testing.
* Injury preventing completion of the intervention.

Ages: 17 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Change in countermovement jump (CMJ) jump height | Baseline and after 8 weeks of intervention.
  Change in vertical jump height (cm) measured with dual force plates during a countermovement jump, from baseline (pre-test) to post-intervention (8 weeks).
Change in Sprint Speed (30 m sprint test using 1080 Sprint system) | Baseline and after 8 weeks of intervention.
  Change in sprint velocity (m/s) and split times (0-5 m, 0-10 m, 0-30 m).
Change in Drop Jump Reactive Strength Index (RSI) | Baseline and after 8 weeks.
  Change in reactive strength index (jump height / ground contact time) measured during drop jump from 30 cm platform.

SECONDARY OUTCOMES:
Change in Standing Broad Jump Distance (SBJ) | Baseline and after 8 weeks.
  Change in Standing Broad Jump Distance (SBJ)
Change in Sprint Mechanics (1080 Sprint) | Baseline and after 8 weeks.
  Change in peak force (N) and peak power (W) during 30 m sprint.
Change in Change-of-Direction Performance (15-0-5 test) | Baseline and after 8 weeks.
  Change in time (s) to complete 15-0-5 change-of-direction test, including deceleration and re-acceleration phases.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Pupiš, Study Chair — Faculty of Sport Science and Health, Matej Bel University; Marián Škorik, Principal Investigator — Faculty of Sport Science and Health, Matej Bel University
Locations (1):
- Masaryk University, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including pre- and post-intervention performance outcomes (e.g., jump height, reactive strength index, sprint performance, change-of-direction test results), will be shared. No personally identifying information will be included. Data will be shared through an open repository such as OSF (Open Science Framework) or Zenodo. The link will be provided upon availability.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data and supporting information will be available beginning 12 months after article publication. Data will remain available for at least 5 years after publication.
Access Criteria: Qualified researchers will be able to request access to the de-identified dataset and supporting materials by contacting the corresponding author. Access will be granted for scientific purposes only and in accordance with institutional and ethical guidelines.

REFERENCES:
- [Background] Afonso J, Nakamura FY, Baptista I, Rendeiro-Pinho G, Brito J, Figueiredo P. Microdosing: Old Wine in a New Bottle? Current State of Affairs and Future Avenues. Int J Sports Physiol Perform. 2022 Oct 6;17(11):1649-1652. doi: 10.1123/ijspp.2022-0291. Print 2022 Nov 1. PMID 36202386
- [Background] Cuadrado-Penafiel V, Castano-Zambudio A, Martinez-Aranda LM, Gonzalez-Hernandez JM, Martin-Acero R, Jimenez-Reyes P. Microdosing Sprint Distribution as an Alternative to Achieve Better Sprint Performance in Field Hockey Players. Sensors (Basel). 2023 Jan 6;23(2):650. doi: 10.3390/s23020650. PMID 36679451
- [Background] Wang J, Wang Y, Jiang Y, Li S, Jia X, Xiao X, Sun W, Wang P, Zhang Q. Datasets-Based IMPDH1 Revisited: Heterozygous Missense Variants for Dominant Retinitis Pigmentosa While Truncation Variants Are Likely Non-Pathogenic. Curr Eye Res. 2024 Aug;49(8):853-861. doi: 10.1080/02713683.2024.2336158. Epub 2024 Apr 11. PMID 38604988
- [Background] DiStefano LJ, Martinez JC, Crowley E, Matteau E, Kerner MS, Boling MC, Nguyen AD, Trojian TH. Maturation and Sex Differences in Neuromuscular Characteristics of Youth Athletes. J Strength Cond Res. 2015 Sep;29(9):2465-73. doi: 10.1519/JSC.0000000000001052. PMID 26313573
- [Background] Liu G, Wang X, Xu Q. Microdosing Plyometric Training Enhances Jumping Performance, Reactive Strength Index, and Acceleration among Youth Soccer Players: A Randomized Controlled Study Design. J Sports Sci Med. 2024 Jun 1;23(2):342-350. doi: 10.52082/jssm.2024.342. eCollection 2024 Jun. PMID 38841635
- [Background] Nuzzo JL, Pinto MD, Kirk BJC, Nosaka K. Resistance Exercise Minimal Dose Strategies for Increasing Muscle Strength in the General Population: an Overview. Sports Med. 2024 May;54(5):1139-1162. doi: 10.1007/s40279-024-02009-0. Epub 2024 Mar 20. PMID 38509414